CLINICAL TRIAL: NCT02298166
Title: Dose-Finding Run-in Phase I Followed by a Phase III, Multicenter, Randomized, Double-Blind, Placebo-controlled Study of Crenolanib in Combination With Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia and Activating FLT3 Mutations
Brief Title: Study of Crenolanib in Combination With Chemotherapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia and Activating FLT3 Mutations
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The manufacturer Arog Pharmaceuticals Inc has terminated the Agreement Concerning the Support of an Investigator Initiated Trial this became valid on 2020/03/09
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMLSG 19-13 / ARO-007
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; FLT3 mutations; Crenolanib; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Drug Therapy; Mitoxantrone; Cytarabine; crenolanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (Placebo Comparator): chemotherapy (MC) in combination with placebo
  Interventions: Drug: chemotherapy (Mitoxantrone, Cytarabine); Drug: Placebo; Other: Allogeneic stem cell transplantation
- Experimental arm (Experimental): chemotherapy (MC) in combination with crenolanib
  Interventions: Drug: chemotherapy (Mitoxantrone, Cytarabine); Drug: Crenolanib; Other: Allogeneic stem cell transplantation

INTERVENTIONS:
Drug: chemotherapy (Mitoxantrone, Cytarabine) — Induction therapy:
  * Mitoxantrone 10 mg/m² IV, push (8 mg/m² for patients > 60 years of age and/or previous allogeneic HCT) d 1-3
  * Cytarabine 1000 mg/m² IV (500 mg/m² for patients > 60 years of age and/or previous allogeneic HCT), over 3 hours, d 1-6
  Consolidation therapy:
  Younger adult patients (18 to 60 yrs):
  Cytarabine 1500 mg/m² by i.v infusion over 3 hours BID on days 1-3 (total dose 9000 mg/m²).
  Older patients (> 60 yrs) and or previous allogeneic HCT:
  Cytarabine 1000 mg/m² by i.v. infusion over 3 hours BID on days 1-3 (total dose 6000 mg/m²).
Drug: Placebo — Induction therapy:
  Placebo to be given as p.o. TID starting d 7+, given continuously thereafter until 48 hours prior to the next chemotherapy.
  Consolidation therapy:
  Placebo will start on day 4, thereafter with continuous dosing until 48h before start of subsequent consolidation chemotherapy.
  Maintenance therapy with placebo is intended in all patients after allogeneic HCT or intermediate-dose cytarabine consolidation therapy. Maintenance therapy will be given for 364 days (equivalent to 13 cycles à 28 days) after recovery from allogeneic HCT or IDAC.
  Maintenance with placebo will be given at the same dose tolerated during induction therapy.
  Arms: Standard arm
Drug: Crenolanib — Induction therapy:
  Crenolanib to be given as p.o. TID starting d 7+, given continuously until 48 hours prior to the next chemotherapy.
  Consolidation therapy:
  Crenolanib will start on day 4, thereafter with continuous dosing until 48h before start of subsequent consolidation chemotherapy.
  Maintenance therapy with Crenolanib is intended in all patients after allogeneic HCT or intermediate-dose cytarabine consolidation therapy. Maintenance therapy will be given for 364 days (equivalent to 13 cycles à 28 days) after recovery from allogeneic HCT or IDAC.
  Maintenance with Crenolanib will be given at the same dose tolerated during induction therapy.
  Arms: Experimental arm
Other: Allogeneic stem cell transplantation — In patients achieving a CR or CRi after salvage-reinduction chemotherapy allogeneic HCT from a matched related or unrelated donor is the preferred form of consolidation. Preferred source of allogeneic HSC are mobilized peripheral blood stem cells. Other forms of allogeneic transplantation (haploidentical donor; cord blood) are allowed.
  Allogeneic HCT should be conducted at the earliest time point after the start of the last chemotherapy but no later than after 56 days. A delay of transplant beyond this time window need to be discussed with the Coordinating Investigator. Patients can receive allogeneic HCT directly after salvage re-induction chemotherapy with MC, but also later on following consolidation with IDAC.

SUMMARY:
The main trial is a double-blinded, placebo-controlled, randomized, phase III, multi-center trial in adult patients with relapsed or refractory AML harboring an activating FLT3 mutation as defined in the inclusion /exclusion criteria.

An initial open label dose-finding run-in phase I of the study will be performed administering the study drug crenolanib with salvage chemotherapy consisting of mitoxantrone and cytarabine (MC) in 18 patients according to the experimental arm of the study. After completion of this dose-finding run-in phase I, toxicity and response data will be provided to the external Data and Safety Monitoring Board (DSMB) and the Trial Committee by the Coordinating Investigator. The Trial Committee will decide on the basis of these data and the recommendation of the DSMB on dose modification and the further conduct of the study with regard to the double-blinded, placebo-controlled, randomized phase of the study.

The double-blinded, placebo-controlled randomized portion will start after the completion of the dose-finding run-in phase I and positive opinion of the Trial Committee.

Crenolanib starts on day 7 of MC and is given continuously until 48 hours prior to the next chemotherapy; if receiving allogeneic HCT, crenolanib is held 48 hours prior to conditioning and restarts no sooner than 30 days and not later than day 100 after transplant.

Sample size randomized phase: 276 patients

Primary objective: To evaluate the impact of crenolanib given in combination with salvage chemotherapy and consolidation including allogeneic hematopoietic cell transplantation and ongoing single agent maintenance therapy with crenolanib on event-free (EFS) and overall survival (OS) in adult patients with relapsed or refractory AML harboring FLT3 activating mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of AML either refractory to induction therapy or relapsed after first line treatment including chemotherapy, autologous and allogeneic HCT

   1. refractory to induction therapy is defined as no CR, CRi, PR (according to standard criteria, 28) after one intensive induction therapy including at least 7 days of cytarabine 100-200mg/m² continuously or an equivalent regimen with cytarabine with total dose not less than 700mg/m² per cycle and 3 days of an anthracycline (e.g. daunorubicin, idarubicin)
   2. relapsed after first line therapy is defined as relapsed AML (according to standard criteria, 28) after a first line therapy including at least one intensive induction and consolidation therapy
2. Presence of FLT3-activating mutation at the time of refractory disease or relapse assessed in the central AMLSG reference laboratory within AMLSG BiO study (ClinicalTrials.gov Identifier: NCT01252485); positivity of FLT3-ITD and FLT3-TKD is defined based on genescan analysis with a mutant to wild-type ratio equal or above 5%
3. Patients considered eligible for intensive chemotherapy
4. ECOG performance status of ≤ 2
5. Age ≥ 18 years with the capacity to give written informed consent
6. Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months).
7. Female patients of reproductive age must agree to avoid getting pregnant while on therapy and for 3 months after the last dose of crenolanib.
8. Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy). Hormonal contraception is an inadequate method of birth control.
9. Men must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 3 month after the last dose of crenolanib).
10. Willing to adhere to protocol specific requirements
11. Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Known or suspected hypersensitivity to the study drugs and/or any excipients
2. ECOG performance status >2
3. Inadequate cardiac, hepatic and/or renal function at the Screening Visit defined as:

   * ejection fraction < 45% confirmed by echocardiography
   * creatinine >1.5x upper normal serum level
   * total bilirubin > upper normal serum level
   * AST or ALT >2x upper normal serum level
4. Active central nervous system involvement
5. Any clinically significant, advanced or unstable disease or history of that may interfere with primary or secondary variable evaluations or put the patient at special risk, such as:

   * Myocardial infarction, unstable angina within 3 months before screening
   * Heart failure NYHA III/IV
   * Severe obstructive or restrictive ventilation disorder
   * Uncontrolled infection
6. Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
7. Currently receiving a therapy not permitted during the study, as defined in Section 10.6.5
8. Active Graft-versus-Host Disease (GvHD) under immunosuppressive therapy different from steroids
9. Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
10. Pre-existing liver disease (e.g.,. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
11. Known history of positive test for hepatitis B surface antigen (HsbAg) or hepatitis C antibody or history of positive test for Human Immunodeficiency Virus (HIV)
12. Hematologic disorder independent of leukemia
13. No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation
14. No consent for biobanking
15. Current participation in any other interventional clinical study within 30 days before the first administration of the investigational product or at any time during the study
16. Patients known or suspected of not being able to comply with this trial protocol
17. Breast feeding women or women with a positive pregnancy test at Screening visit
18. Patients of childbearing potential not willing to use adequate contraception during study and 3 months after last dose of crenolanib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Event-free Survival (EFS) | 4 years
Overall Survival (OS) | 4 years

SECONDARY OUTCOMES:
Rates of complete remission (CR) and complete remission with incomplete blood count recovery (CRi) after induction therapy | 2 months
Cumulative incidence of relapse (CIR) | 4 years
Cumulative incidence of death (CID) | 4 years
Quality of life (QoL) | 5.5 years
  Quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, and demographics (24) at the Screening visit, after last induction cycle, after last consolidation cycle, at end of treatment visit and every year thereafter.
Rate of early deaths or hypoplastic deaths (ED or HD) | 2 months
Toxicity: Type, frequency, severity, timing and relatedness of hematologic and non-hematologic toxicities | 1.5 years
  Type, frequency, severity, timing and relatedness of hematologic and non-hematologic toxicities

CONTACTS AND LOCATIONS:
Locations (1):
- Ulm University Hospital, Ulm, Germany